CLINICAL TRIAL: NCT05502237
Title: A Randomized, Open-Label, Phase 3 Study to Evaluate Zimberelimab and Domvanalimab in Combination With Chemotherapy Versus Pembrolizumab With Chemotherapy for the First-Line Treatment of Patients With Metastatic Non-Small Cell Lung Cancer With No Epidermal Growth Factor Receptor or Anaplastic Lymphoma Kinase Genomic Tumor Aberrations
Brief Title: Zimberelimab and Domvanalimab in Combination With Chemotherapy Versus Pembrolizumab With Chemotherapy in Patients With Untreated Metastatic Non-Small Cell Lung Cancer
Acronym: STAR-121
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Collaborators: Arcus Biosciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GS-US-626-6216; 2022-000578-25 (EudraCT Number)
Record Dates: First submitted 2022-08-12; First posted 2022-08-16 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — zimberelimab; pembrolizumab; Carboplatin; Cisplatin; Paclitaxel; 130-nm albumin-bound paclitaxel; Pemetrexed

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Zimberelimab (ZIM) +Domvanalimab (DOM) + Chemotherapy (Experimental): Participants will receive ZIM 360 mg + DOM 1200 mg (up to 35 doses) with chemotherapy every 3 weeks (Q3W) on Day 1 of each 21-day cycle.
  Choice of chemotherapy is dependent on histology.
  * Participants with nonsquamous histology will receive cisplatin 75 mg/m^2 or carboplatin area under the concentration versus time curve (AUC)5 + pemetrexed 500 mg/m^2 Q3W for first 4 cycles. After the completion of the first 4 cycles, participants with nonsquamous histology may continue with maintenance pemetrexed 500 mg/m^2 Q3W until disease progression or intolerable toxicities.
  * Participants with squamous histology will receive carboplatin AUC 6 Q3W with paclitaxel 200 mg/m^2 Q3W or nab-paclitaxel 100 mg/m^2 weekly (QW) for first 4 cycles.
  Interventions: Drug: Zimberelimab; Drug: Domvanalimab; Drug: Carboplatin; Drug: Cisplatin; Drug: Paclitaxel; Drug: Nab-paclitaxel; Drug: Pemetrexed
- Pembrolizumab (PEMBRO) + Chemotherapy (Active Comparator): Participants will receive PEMBRO 200 mg (up to 35 doses) with chemotherapy Q3W on Day 1 of each 21-day cycle.
  Choice of chemotherapy is dependent on histology.
  * Participants with nonsquamous histology will receive cisplatin 75 mg/m^2 or carboplatin AUC 5 + pemetrexed 500 mg/m^2 Q3W for first 4 cycles. After the completion of the first 4 cycles, participants with nonsquamous histology may continue with maintenance pemetrexed 500 mg/m^2 Q3W until disease progression or intolerable toxicities.
  * Participants with squamous histology will receive carboplatin AUC 6 Q3W with paclitaxel 200 mg/m^2 Q3W or nab-paclitaxel 100 mg/m^2 weekly (QW) for first 4 cycles.
  Interventions: Drug: Pembrolizumab; Drug: Carboplatin; Drug: Cisplatin; Drug: Paclitaxel; Drug: Nab-paclitaxel; Drug: Pemetrexed
- Zimberelimab (ZIM) + Chemotherapy (Experimental): Participants will receive ZIM 360 mg (up to 35 doses) with chemotherapy Q3W on Day 1 of each 21-day cycle.
  Choice of chemotherapy is dependent on histology.
  * Participants with nonsquamous histology will receive cisplatin 75 mg/m^2 or carboplatin AUC 5 + pemetrexed 500 mg/m^2 Q3W for first 4 cycles After the completion of the first 4 cycles, participants with nonsquamous histology may continue with maintenance pemetrexed 500 mg/m^2 Q3W until disease progression or intolerable toxicities.
  * Participants with squamous histology will receive carboplatin AUC 6 Q3W with paclitaxel 200 mg/m^2 Q3W or nab-paclitaxel 100 mg/m^2 weekly (QW) for first 4 cycles.
  Interventions: Drug: Zimberelimab; Drug: Carboplatin; Drug: Cisplatin; Drug: Paclitaxel; Drug: Nab-paclitaxel; Drug: Pemetrexed

INTERVENTIONS:
Drug: Zimberelimab — Administered intravenously
  Other Names: GS-0122; AB122
  Arms: Zimberelimab (ZIM) + Chemotherapy; Zimberelimab (ZIM) +Domvanalimab (DOM) + Chemotherapy
Drug: Domvanalimab — Administered intravenously
  Other Names: GS-0154; AB154
  Arms: Zimberelimab (ZIM) +Domvanalimab (DOM) + Chemotherapy
Drug: Pembrolizumab — Administered intravenously
  Other Names: KEYTRUDA®
  Arms: Pembrolizumab (PEMBRO) + Chemotherapy
Drug: Carboplatin — Administered intravenously
Drug: Cisplatin — Administered intravenously
Drug: Paclitaxel — Administered intravenously
Drug: Nab-paclitaxel — Administered intravenously
Drug: Pemetrexed — Administered intravenously

SUMMARY:
The primary objective of this study is to compare the effect of zimberelimab (ZIM) and domvanalimab (DOM) in combination with chemotherapy relative to pembrolizumab (PEMBRO) in combination with chemotherapy on overall survival (OS) in patients with untreated metastatic non-small cell lung cancer with no actionable genomic alteration.

ELIGIBILITY:
Key Inclusion Criteria:

* Life expectancy ≥ 3 months.
* Pathologically documented NSCLC that meets both of the criteria below:

  * Have documented evidence of Stage IV NSCLC disease at the time of enrollment (based on American Joint Committee on Cancer (AJCC), Eighth Edition).
  * Have documented negative test results for epidermal growth factor receptor (EGFR) and anaplastic lymphoma kinase (ALK) mutations.
* Have no actionable genomic alterations such as ROS proto-oncogene 1 (ROS1), neurotrophic tyrosine receptor kinase (NTRK), proto-oncogene B-raf (BRAF), RET mutations, or other driver oncogenes with approved frontline therapies.
* Have not received prior systemic treatment for metastatic NSCLC.
* Measurable disease per RECIST v1.1 criteria by investigator assessment.
* Eastern Cooperative Oncology Group performance status (ECOG PS) score of 0 or 1.
* Have adequate organ functions.

Key Exclusion Criteria:

* Have mixed small-cell lung cancer (SCLC) and NSCLC histology.
* Positive serum pregnancy test or individuals who are breastfeeding or have plans to breastfeed during the study period.
* Received prior treatment with any anti-PD-1, anti-PD-L1, or any other antibody targeting an immune checkpoint.
* Known hypersensitivity to the study drug, its metabolites, or formulation excipient.
* Have an active second malignancy or have had an active second malignancy within 3 years prior to enrollment.
* Have an active autoimmune disease that required systemic treatment in past 2 years (i.e., with use of disease-modifying agents, corticosteroids, or immunosuppressive drugs).
* Are receiving chronic systemic steroids.
* Have significant third-space fluid retention.
* Have untreated central nervous system (CNS) metastases and/or carcinomatous meningitis.
* Active chronic inflammatory bowel disease (ulcerative colitis, Crohn's disease) or gastrointestinal perforation within 6 months of enrollment.
* Has a history of (noninfectious) pneumonitis/interstitial lung disease that required steroids or has current pneumonitis/interstitial lung disease.
* Has had an allogenic tissue/solid organ transplant.
* Have received a live-virus vaccination within 30 days of planned treatment start. Seasonal flu and COVID-19 vaccines that do not contain live virus are permitted.
* Have known active hepatitis B virus (HBV) or hepatitis C virus (HCV) infection.

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1021 (Actual)
Dates: Start 2022-10-12 (Actual); Primary Completion 2028-06 (Estimated); Study Completion 2029-01 (Estimated)

PRIMARY OUTCOMES:
Overall Survival (OS) in Participants With Positive Programmed Cell Death-Ligand 1 (PD-L1) Expression (≥1%Tumor Cells) and in all Randomized Participants. | Up to 68 months
  OS is defined as the time from the date of randomization to the date of death from any cause.

SECONDARY OUTCOMES:
Progression-free Survival (PFS) as Assessed by Blinded Independent Central Review (BICR) per Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1 | Upt to 50 months
  PFS is defined as the time from the date of randomization until disease progression (PD) or death from any cause, whichever comes first.
Objective Response Rate (ORR) as Assessed by BICR per RECIST Version 1.1 | Up to 50 Months
  ORR is defined as the proportion of participants who have achieved a complete response (CR) or partial response (PR) that is confirmed at least 4 weeks later.
Duration of Response (DOR) as Assessed by BICR per RECIST Version 1.1 | Up to 50 Months
  DOR is defined as the time from the first response (CR or PR), to the first documented PD or death from any cause, whichever comes first.
Percentage of Participants Experiencing Treatment-emergent Adverse Events (TEAEs) | First dose date up to 50 months plus 30 days
Percentage of Participants Experiencing Clinical Laboratory Abnormalities | First dose date up to 50 months plus 30 days
Time to First Symptom Deterioration in Non-small Cell Lung Cancer Symptom Assessment Questionnaire (NSCLC-SAQ) Total Score | Baseline, Up to 50 Months
  The NSCLC-SAQ is a patient reported outcome measure with seven items assessing five symptom concepts of NSCLC: cough, pain, dyspnea, fatigue, and appetite. Each item is rated using a five-point verbal rating scale from "No <symptom> At All" to "Very severe <symptom>" or from "Never to Always," corresponding to a score of 0 to 4. The sum of all 5 domain scores will be computed, if any scores are missing, a total score will not be computed. The total score ranges between 0 and 20 with higher scores indicating more severe symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (186):
- United States (11):
  - Innovative Clinical Research Institute, Whittier, California
  - George Washington Medical Faculty Associates, Washington D.C., District of Columbia
  - Moffitt Cancer Center, Tampa, Florida
  - Illinois Cancer Care, Peoria, Illinois
  - Messino Cancer Centers, Asheville, North Carolina
  - Oncology Hematology Care, Inc., Cincinnati, Ohio
  - Hematology & Oncology Associates, Eugene, Oregon
  - AHN Allegheny General Hospital, Pittsburgh, Pennsylvania
  - Texas Oncology - Austin, Austin, Texas
  - Oncology and Hematology Associates of Southwest Virginia, Inc, Blacksburg, Virginia
  - Northwest Cancer Specialists, PC, Vancouver, Washington
- Argentina (8):
  - Investigaciones CORI S.R.L., Capital
  - Centro Médico Privado Centro de Especialidades Médicas Ambulatorias e Investigación Clínica, Cardoba
  - Sanatorio Allende, Córdoba
  - Sanatorio Britanico de Rosario, Rosario
  - Sanatorio Parque de Rosario, Rosario
  - Hospital Provincial del Centenario, Rosario
  - Instituto Medico de la Fundacion Estudios Clinicos, Rosario
  - Clínica Viedma, Viedma
- Austria (3):
  - Ordensklinikum Linz GmbH, Elisabethinen, Linz
  - Krankenhaus Nord - Klinik Floridsdorf, Vienna
  - Klinikum Wels-Grieskirchen, Wels
- Belgium (4):
  - Algemeen Ziekenhuis Sint-Lucas, Aalst
  - Grand Hopital de Charleroi asbl (GHdC), Charleroi
  - AZ Sint-Maarten, Mechelen
  - CHU UCL Namur / Site Sainte Elisabeth, Namur
- Brazil (11):
  - Cenantron Centro Avançado de Tratamento Oncologico Ltda, Belo Horizonte
  - Hospital Evangelico de Cachoeiro de Itapemirim, Cachoeiro de Itapemirim
  - Fundacao Universidade De Caxias Do Sul - FUCS/RS, Caxias do Sul
  - Instituto do Câncer do Ceará - ICC, Fortaleza
  - Oncosite - Centro de Pesquisa Clinica em Oncologia LTDA, Ijuí
  - Irmandade da Santa Casa de Misericordia de Porto Alegre, Porto Alegre
  - Hospital de Clínicas de Porto Alegre, Porto Alegre
  - Hospital São Lucas da PUCRS, Porto Alegre
  - Hospital Ana Nery Santa Cruz do Sul, Santa Cruz do Sul
  - Instituto Brasiliero de Controle do Cancer IBCC, São Paulo
  - Centro Des Pesquisas Clinicas da Fundacao Doutor Amaral Carvalho, São Paulo
- Canada (4):
  - Centre Integre de sante et de services sociaux de la Monteregie Centre, Greenfield Park
  - Moncton Hospital, Moncton
  - CISSS des Laurentides, Québec
  - Centre de santé et services sociaux de Rimouski-Neigette, Rimouski
- Chile (7):
  - Clinica Alemana de Santiago, Las Condes
  - Clinica Puerto Montt, Port Montt
  - Orlandioncologia, Providencia
  - Oncovida- Santiago, Providencia
  - Biocinetic, Santiago
  - James Lind Centro de Investigacion del Cancer, Temuco
  - Oncocentro APYS, Viña del Mar
- China (22):
  - West China Hospital Sichuan University, Chengdu
  - Chongqing University Cancer Hospital, Chongqing
  - Deyang People's Hospital, Deyang
  - Fujian Cancer Hospital, Fuzhou
  - The First Affiliated Hospital of Guangzhou Medical University, Guangzhou
  - Guangzhou First People's Hospital, Guangzhou
  - Zhejiang Cancer Hospital, Hangzhou
  - The Second Affiliated Hospital of Nanchang University, Jiangxi
  - Shandong Cancer Hospital, Jinan
  - Jiangxi Chest Hospital, Nanchang
  - Nanjing Drum Tower Hospital, Nanjing
  - Guangxi Medical University Cancer Hospital, Nanning
  - Shanghai Chest Hospital, Shanghai
  - Shanghai East Hospital, Shanghai
  - Shanghai Pulmonary Hospital, Shanghai
  - Cancer Hospital of Shantou University Medical College, Shantou
  - Tianjin Medical University Cancer Institute & Hospital, Tianjin
  - Union Hospital Tongji Medical College Huazhong University of Science and Technology, Wuhan
  - Tongji Hospital Tongji Medical College of Hust, Wuhan
  - The First Affiliated Hospital of Xian Jiaotong University, Xi'an
  - The First Affiliated Hospital of Xinxiang Medical College, Xinxiang
  - Henan Cancer Hospital, Zhengzhou
- France (9):
  - Ambroise-Pare Hospital, Assistance Publique - Hopitaux de Paris, Boulogne-Billancourt
  - Clinique Victor Hugo, Centre de Cancerologie de la Sarthe, Le Mans
  - Hopital Nord, Marseille
  - Institut de Cancer de Montpellier (ICM) - Val d'Aurelle, Montpellier
  - Institut de cancerologie de l'ouest (ICO), Saint-Herblain
  - Hopital d'Instruction des Armees (HIA) Begin, Saint-Mandé
  - Centre Hospitalier de Saint-Quentin, Saint-Quentin
  - Hôpital Foch, Suresnes
  - CHI de Toulon la Seyne-sur-Mer Hopital Sainte Musse, Toulon
- Germany (11):
  - Kliniken der Stadt Köln ggmbh, Krankenhaus Koln-Merheim/Lungenklinik, Cologne
  - Universitatsklinikum Essen / Westdeutsches Tumorzentrum, Innere Klinik (Tumorforschung), Essen
  - LungenClinic Grosshansdorf, Großhansdorf
  - Krankenhaus Martha-Maria Halle Dölau, Halle
  - Asklepios Kliniken Hamburg, Hamburg
  - Katholisches Marienkrankenhaus gGmbH, Hamburg
  - Lungenklinik Hemer, Zentrum fur Pneumologie and Thoraxchirurgie, Hemer
  - Vincentius-Diakonissen-Kliniken gAG, St. Vincentius-Kliniken, Medizinische Klinik 2, Karlsruhe
  - Universitatsklinikum Schleswig-Holstein, Lübeck
  - Johannes Wesling Klinikum Minden, Minden
  - Sana Klinikum Offenbach GmbH, Medizinische Klinik IV, Hämatologie und Internistische Onkologie, Offenbach
- Hong Kong (3):
  - Queen Elizabeth Hospital, Hong Kong
  - Queen Mary Hospital, Hong Kong
  - Prince of Wales Hospital, New Territories
- Israel (4):
  - Shaare Zedek Medical Center, Jerusalem
  - Oncology Institute, Galilee Medical Center, Route 89 Nahariya-Cabri, Nahariya
  - Rabin Medical Center, Petah Tikva
  - Tel-Aviv Sourasky Medical Center, Tel Aviv
- Italy (10):
  - Azienda Ospedaliera San Giuseppe Moscati, Avellino
  - Azienda Socio Sanitaria Territoriale di Cremona, Cremona
  - Ospedale Policlinico San Martino, Genova
  - Ospedale San Raffaele, Milan
  - AORN Cardarelli, Naples
  - IRCCS Policlinico S. Matteo, Dipartimento Oncologia Ematologia-Oncologia Medica, Pavia
  - Azienda Sanitaria Territoriale Pesaro e Urbino (AST), Pesaro
  - Ospedale Guglielmo da Saliceto AUSL di Piacenza, Piacenza
  - Centro di Riferimento Oncologico, Pordenone
  - Regina Elena Institute for Cancer Research, Rome
- Japan (15):
  - National Cancer Center Hospital East, Chiba
  - National Hospital Organization Shikoku Cancer Center, Ehime
  - Kyushu University Hospital, Fukuoka
  - Kurume University Hospital, Fukuoka
  - National Hospital Organization Himeji Medical Center, Hyōgo
  - Hyogo Cancer Center, Hyōgo
  - Kanazawa University Hospital, Ishikawa
  - Kanagawa Cancer Center, Kanagawa
  - Sendai Kousei Hospital, Miyagi
  - Niigata Cancer Center Hospital, Niigata
  - Osaka Metropolitan University Hospital, Osaka
  - Osaka Medical and Pharmaceutical University Hospital, Osaka
  - Kindai University Hospital, Osaka
  - National Hospital Organization Kinki Chuo Chest Medical Center, Osaka
  - Saitama Medical University, Saitama
- Mexico (7):
  - Health Pharma Professional Research S.A. de C.V., México
  - Hospital Universitario Dr. Jose Eleuterio Gonzalez, Mitras Centro
  - Oaxaca Site Management Organization, Oaxaca City
  - Centro de Investigacion Clinica de Oaxaca, Oaxaca City
  - Clinical Medical Research SC., Orizaba Centro
  - Clinica Integral Internacional de Oncologia S de RL de CV, Puebla City
  - FAICIC Clínical Research, Veracruz
- Netherlands (5):
  - Amphia Ziekenhuis, Breda
  - Ziekenhuis Gelderse Vallei, Ede
  - Universitair Medisch Centrum Groningen, Groningen
  - Ziekenhuis St Jansdal, Harderwijk
  - TweeSteden Ziekenhuis, Tilburg
- Portugal (6):
  - Hospital Prof. Doutor Fernando Fonseca, Amadora
  - Instituto Português de Oncologia de Lisboa Francisco Gentil, Lisbon
  - Fundacao Champalimaud, Lisbon
  - Hospital Beatriz Angelo. Hospital de Loures., Lisbon
  - Centro Hospitalar Universitário Lisboa Norte - Hospital Pulido Valente, Lisbon
  - Unidade Local de Saude de Matosinhos EPE - Hospital Pedro Hispano SA, Senhora da Hora
- Tang Tock Seng Hospital, Singapore, Singapore
- South Korea (7):
  - Samsung Medical Center, Gangnam-Gu
  - National Cancer Center, Goyang
  - Chungbuk National University Hospital, Heungdeok-Gu
  - Gachon University Gil Medical Center, Inchon
  - Severance Hospital, Yonsei University Health System, Seoul
  - The Catholic University of Korea, Seoul St. Mary's Hospital, Seoul
  - The Catholic University of Korea, Saint Vincent's Hospital, Suwon
- Spain (20):
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital de la Santa Creu i de Sant Pau, Barcelona
  - Hospital Universitari Dexeus (USP Institut Universitari Dexeus/Hospital Universitari Quiron Dexeus), Barcelona
  - Hospital Universitari Vall D'Hebron, Barcelona
  - Hospital Parc Tauli, Barcelona
  - Hospital Universitario Reina Sofia, Córdoba
  - Hospital Doctor Josep Trueta, Girona
  - Hospital Universitario de Jaen, Jaén
  - Hospital Universitario de Canarias, Las Palmas de Gran Canaria
  - Hospital Universitario Fundacion Jimenez Diaz, Madrid
  - Clinica Universidad de Navarra, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario Puerta de Hierro de Majadahonda, Majadahonda
  - Hospital Sant Joan de Reus, Reus
  - Hospital Regional Universitario de Malaga, Rincón de la Victoria
  - Hospital Universitario Virgen Macarena, Seville
  - Hospital Universitario Virgen del Rocio, Seville
  - Instituto Valenciano De Oncologia (IVO), Valencia
  - Hospital Universitari i Politecnic La Fe, Valencia
  - Hospital Vithas Valencia 9 de Octubre, Valencia
- Taiwan (8):
  - Changhua Christian Hospital, Changhua
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - E-DA Hospital, Kaohsiung City
  - Chang Gung Memorial Hospital Kaohsiung, Kaohsiung City
  - Chi Mei Hospital, Liouying, Tainan
  - Taipei Veterans General Hospital, Taipei
  - National Taiwan University Hospital, Taipei
  - Chang Gung Memorial Hospital Linkou Branch of the Chang Gung Medical Foundation, Taoyuan
- Turkey (Türkiye) (8):
  - Ankara Bilkent Sehir Hastanesi, Ankara
  - Dr. Abdurrahman Yurtaslan Ankara Onkoloji Egitim ve Arastirma Hastanesi, Ankara
  - Trakya University Faculty of Medicine, Edirne
  - Istanbul University Cerrahpasa Medical Faculty Hospital, Fatih
  - Goztepe Prof. Dr. Suleyman Yalcın Sehir Hastanesi, Istanbul
  - Medipol Mega University Hospital, Istanbul
  - Acibadem Mehmet Ali Aydinlar Universitesi Atakent Hastanesi, Kaakaekmece
  - Turgut Ozal Medical Faculty, Malatya
- United Kingdom (2):
  - St Bartholomew's Hospital, Barts Health NHS Trust, London
  - The Christie NHS Foundation Trust, Department of Medical Oncology, Manchester

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Gilead Clinical Trials Website — https://www.gileadclinicaltrials.com/study/?id=GS-US-626-6216